CLINICAL TRIAL: NCT05342935
Title: A Prospective, Open-label, Cross-over, Multi-center Pilot Study to Evaluate the Safety, Feasibility and Usability of the IDA in Subjects Suffering From a Stage 5 Kidney Disease and Who Are Treated With Peritoneal Dialysis
Brief Title: A Prospective, Open-label, Multi-center Pilot Study to Evaluate the Safety, Feasibility and Usability of the IDA
Acronym: CSP-027-21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: liberDi Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: liberDi
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease Stage V

STUDY DESIGN:
Intervention Model Description: Subjects will pursue their usual manual PD exchanges, followed by the treatment with the investigational device and then back to their manual PD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IDA treatment (Experimental): Each subject will be treated with his prescribed manual PD for 14 days, followed by a treatment period of 14 days with the investigational IDA system, and concluding with additional 14 days of treatment with the manual PD.
  Interventions: Device: Inteligent Dialysis Assistant (IDA)

INTERVENTIONS:
Device: Inteligent Dialysis Assistant (IDA) — The IDA is a small dialysis system that allows a higher level of freedom to the patients, permitting them to perform the PD exchange while continuing to do their everyday activities

SUMMARY:
This is a multi-center, open label, cross-over clinical study. A total of 15 subjects will be enrolled to use the IDA for every peritoneal dialysis exchange for 14 days. To participate in the study, the subjects must have current CKD5 and have been treated with PD for at least 3 months. The subjects will undergo a single peritoneal dialysis exchange procedure at the PD clinic, under supervision of the medical staff and instructed about its operation. Further exchanges will be performed by the subjects themselves at home.

The study includes three periods:

First period (Observational): 14-day Observational Period. Eligible subjects who sign informed consent will continue with their regular CAPD treatment while performing measurement and recording of dialysate in/out time.

Second period (Interventional): 14-day interventional period, where subjects will perform dialysis exchanges using the IDA according to the below visit schedule.

Third period (Follow up): 14-day follow up period, during which the study staff will call the subject once weekly to inquire about device-related SAEs and any changes to concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CKD stage 5 under peritoneal dialysis
* Age ≥18 years
* Mental ability to understand the study procedures and provide informed consent
* At least 3 months on peritoneal dialysis prior to enrollment
* At least 3 daily exchanges
* Stable PD prescription for the last 2 months
* Subject who is self-treated

Exclusion Criteria:

* Need of cycler (APD)
* Known Mechanical problem during the last month (i.e. drainage or fill problems)
* Pregnant or breastfeeding women, and women with childbearing potential who is unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the entire clinical trial period.
* Subjects who are unwilling or unable to comply with study procedures
* Known Peritonitis or other catheter related infection during the last 3 months prior to enrollment
* Known Congestive Heart Failure stage III-IV
* Any history of kidney malignancy
* Any planned hospitalization for elective Procedure(s)throughout the duration of participation in the study
* Non-elective hospitalization in the last 3 months prior to enrollment
* Any other medical or mental condition, that at the investigator's discretion may prevent the subject from participating in the study
* Participation in any other clinical study within 4 weeks prior to enrollment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint - Serious Adverse Events Rate | 42 days
  The safety of the IDA, as determined by the accumulative incidence of device-related SAEs throughout the 14-day prospective study period

SECONDARY OUTCOMES:
IDA Usability by Investigator | 14 days
  The usability of the IDA will be evaluated by completing an internal usability questionnaire by the investigator that will check the operation of the various system controls and the ease of use
IDA Usability by Subject | 14 days
  The completion of the internal Satisfaction and QoL internal questionnaire by each participating subject. Answers in the questionnaire range from 1 (poor) to 5 (excellent), and the results range from 6-30 - the higher the result, the higher the subject's wellbeing.
IDA Feasibility | 14 days
  The feasibility of the treatment will be evaluated by recording time length of the in/out PD exchange procedure

CONTACTS AND LOCATIONS:
Overall Officials: Richard Corbett, MD, Principal Investigator — Imperial College Medical Center